CLINICAL TRIAL: NCT01751100
Title: Building Bridges: Addressing HIV Stigma in At-Risk Groups in Community Pharmacies
Brief Title: The Feasibility of Using a General Health Screen to Increase HIV Testing in Community Pharmacies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not receive proper funding to complete this study.
Sponsor: North Bronx Healthcare Network (Other)
Responsible Party: Principal Investigator, Yvette Calderon,MD, MS, Professor of Clinical Emergency Medicine, North Bronx Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RFA-MH-13-092-001
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV Test Offer (Active Comparator): Group 1 (Control) is the current standard of care in HIV testing. A trained counselor provides required information to obtain informed consent for HIV testing and provides rapid HIV testing on site.
  Interventions: Behavioral: HIV Test Offer
- General Health Screen Offer (Experimental): In Group 2 (Intervention), a free general health screening is offered that may include a blood pressure check, blood glucose measurement, a Hepatitis C (HCV) test, and an HIV test.
  Interventions: Behavioral: General Health Screen Offer

INTERVENTIONS:
Behavioral: HIV Test Offer — HIV education and counseling from a trained Research Assistant and offering of a free rapid, oral HIV test
  Arms: HIV Test Offer
Behavioral: General Health Screen Offer — A Research Assistant (RA) will provide health education on diabetes, hypertension, and HIV. The RA will then offer free blood pressure check, blood glucose measuring, rapid Hepatitis C (HCV) test, and a free, rapid oral HIV test.
  Arms: General Health Screen Offer

SUMMARY:
The purpose of this study is to see if offering a general health screening tailored towards high-risk groups (African immigrants, injection drug users (IDUs), and minority men who have sex with men (MSM)) will increase human immunodeficiency virus (HIV) testing, counseling, and linkage acceptance rates in community pharmacies.

DETAILED DESCRIPTION:
About one-fifth of HIV-positive people in the United States remain unaware of their HIV status, and these individuals account for the majority of new transmissions. The preponderance of barriers to HIV has delayed diagnoses and treatment for HIV-infected individuals in the US, and such late diagnoses result in poorer outcomes for HIV-infected individuals and increased cost of medical care. The National HIV/AIDS Strategy for the United States has called for expanded HIV testing, but if the investigators simply replicate existing models, the investigators will continue to fail to reach and engage strategic at-risk populations. Project Building Bridges will use a community setting - the pharmacy - to establish an alternative site for HIV testing to engage large numbers of at risk populations, specifically men who have sex with men (MSM) of color, injection drug users (IDU), and African immigrants; increase HIV awareness, and reduce stigma by placing HIV testing in the context of a general health screening. There are two specific aims: 1) Build partnerships with community stakeholders to understand current barriers to HIV testing, and 2) Determine the effectiveness of a health screening approach by measuring acceptance of HIV testing. In the qualitative research phase, we will conduct focus group discussions of MSM of color, IDUs, and African immigrants, led by the Latino Commission on AIDS, a community-based organization with extensive experience in cultural competency training and utilizations of community social networks, especially with higher risk minority populations, to obtain insights that will help increase participation in HIV testing. Data obtained through qualitative work will guide the development of the "health screening" model, which would include other screening tests (like sugar, blood pressure, hepatitis C, etc) with an HIV test, depending on what the high risk groups preferred in the wellness bundle. The hypothesis is that, by tailoring the health screens, this bundling model will circumvent the stigma associated with HIV testing in these high-risk populations and increase HIV testing acceptance rates. The investigators will conduct a two-group randomized control trial comparing the "health screening" model (intervention) to an HIV test offer (control) in community pharmacies in the Bronx. The trial will help determine the preliminary impact on the acceptance of HIV testing when coupled with an overall health wellness screen. The investigators will also conduct a secondary analysis on HIV testing acceptance rates based on each high-risk groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 64 at time of recruitment

Exclusion Criteria:

* Known to be HIV positive
* Unable to understand the consent process for the study; or otherwise unable to consent to HIV testing

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2016-05 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Acceptance of HIV Testing | 30 minutes
  Rate of participation in voluntary rapid oral HIV test in each group

SECONDARY OUTCOMES:
Proportion of African immigrants that accept HIV testing | 30 minutes
  Rate of HIV acceptance among the subgroup African immigrants, comparing between treatment and control groups
Proportion of IDU that accept HIV testing | 30 minutes
  Rate of HIV acceptance among the subgroup IDUs, comparing between treatment and control groups
Proportion of minority MSM that accept HIV testing | 30 minutes
  Rate of HIV acceptance among the subgroup minority MSM, comparing between treatment and control groups
Linkage to Care | up to one year
  Proportion of positively-screened participants that attend follow-up specialized medical care

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Calderon, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States